CLINICAL TRIAL: NCT03429777
Title: Validation of a Smartphone-Based Hearing-in-Noise Test (HearMe)
Acronym: HearMe
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of novelty of study
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Kasra Zarei, Student, University of Iowa
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 201712793
Record Dates: First submitted 2018-01-19; First posted 2018-02-12 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Hearing Loss; Hearing Disorders; Hearing Abnormality; Hearing Disability; Tinnitus
Keywords: Smartphone; Medical application; Hearing-in-noise test; Digits-in-noise test; Speech reception threshold; Hearing Loss; Hearing Disorders; Hearing Abnormalities; Tinnitus; Hearing aids; Cochlear implants
MeSH Terms: conditions — Hearing Loss; Hearing Disorders; Tinnitus

STUDY DESIGN:
Intervention Model Description: For this study the investigators will test at least 50 subjects with some form or hearing loss and 50 control subjects between the ages of 18-80. The subjects will be invited to take the app. The approach for this study is to characterize hearing-in-noise thresholds (also referred to as a speech-reception threshold) as measured by the app in both subject groups.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hearing Loss Group (Experimental): The investigators will characterize hearing-in-noise thresholds (also referred to as a speech-reception threshold) as measured by the HearMe app in patients with hearing loss.
  Interventions: Device: HearMe Smartphone Application
- Control Group (Active Comparator): The investigators will characterize hearing-in-noise thresholds (also referred to as a speech-reception threshold) as measured by the HearMe app in control subjects without any prior or current hearing loss.
  Interventions: Device: HearMe Smartphone Application

INTERVENTIONS:
Device: HearMe Smartphone Application — The HearMe smartphone application is a digits-in-noise test that can be used to digitally quantify speech reception thresholds.
  Other Names: HearMe; HearMe IA

SUMMARY:
The purpose of this project is to validate a quick, easy-to-use and administer smartphone hearing-in-noise test. The Hearing-in-Noise Test (HINT) measures an individual's ability to hear speech in quiet and in noise. HINTs are traditionally done testing both ears together as binaural hearing ability is key in noisy settings and everyday, functional hearing.

The app (called HearMe) can potentially be used to easily and quickly collect hearing-in-noise and speech-in-noise measurements. The smartphone app developed is a hearing-in-noise test that presents the subject with a series of stimuli consisting of a spoken three-digit sequence presented at a varying hearing-to-noise ratio. For each stimulus presentation, the user tap the three-digit sequence. The duration of the app is less than 3 minutes. For this project the investigators will test at least 50 subjects with hearing loss and 50 control subjects between the ages of 18-80. The subjects will be invited to take the app. The approach for this pilot study is to characterize hearing-in-noise thresholds (also referred to as a speech-reception threshold) as measured by the app in both subject groups, and relate it to the phenotype of each group as a preliminary evaluation of the app as well as a preliminary validation against their routinely collected measurements of hearing function (pure-tone audiometry thresholds).

The study will assess the validity of the test construct in measuring hearing-in-noise thresholds, and serve as a foundation for further iterative designs of the app and future validation and characterization studies. This study seeks to validate a developed smartphone HINT on an initial cohort of patients and controls. It is anticipated that patients with hearing loss will display higher signal-to-noise ratio thresholds (as measured by the iPhone app) compared to controls.

DETAILED DESCRIPTION:
Age-related hearing loss, or presbycusis, is highly prevalent among the elderly. It can have a major impact on the quality of life due to progressive communication difficulties that may lead to psychosocial dysfunction and in extreme cases to social isolation and depression. Hearing aids and cochlear implants have evolved rapidly over the past decades and may strongly improve quality of life in elderly with hearing loss. Nevertheless, it is estimated that in the US and Europe only one out of five to six people with substantial hearing loss is actually using hearing aids. In fact, nearly 50% of people with hearing loss never underwent a hearing test at all. This may be due to denial of illness associated with aging or to disbelieve in bene t from hearing aids or cochlear implants. Hearing screening could increase awareness of hearing loss among elderly and identify those who might bene t from amplification. However, classical audiometry (i.e. pure- tone thresholds and speech-recognition in quiet) is not ideal for screening purposes as it is time consuming and it requires expensive equipment including a soundproof booth and a calibrated audiometer.

Over the past decades, several Speech-In-Noise tests were developed to get a better assessment of a person's hearing ability in real-life situations. These tests generally measure the speech reception threshold (SRT) in dB signal to noise ratio (SNR). SRT is determined as the difference between the level of presented speech and background noise at which the tested per- son can correctly reproduce 50% of words or sentences. It is now generally recognized that the SRT is more representative of a patient's hearing ability in real-life situations than pure- tone audiometry or speech recognition in quiet. The Speech- In-Noise test, based on spoken sentences, is still being used in clinical practice. However, its general use for a broad clinical population has been disputed because not every person is able to understand and repeat complete sentences in noise, regardless of his hearing loss. This test is there- fore considered as an assessment of the entire auditory system, including memory and certain linguistic aspects, rather than of hearing loss alone.

In 2013, the Digits-In-Noise (DIN) test was developed, overcoming several shortcomings of the previous telephone test. It uses, for example, wideband signals instead of the limited telephone bandwidth and concatenating digits, spoken by a male voice. The DIN test requires listeners to repeat three spoken numbers (a so-called digit triplet) presented through a headphone, while a continuous noise is presented synchronously to the same ear. The response is then scored correct or incorrect automatically by the computer. Depending on the test setting, the response can either be imputed by the listener him- self or by an administrator. By using simple digits in a closed set paradigm, the contribution of top-down processing and thus the influence of cognitive status is thought to be minimized. For this test, no learning effect was detected, low measurement errors were reported (0.7 dB SNR for normal-hearing listeners) and high validity was claimed by comparing measured digit- triplet SRTs and sentence SRTs. Although SRT-in-noise reflects different aspects of hearing acuity than pure-tone thresholds, both measures are also highly correlated. Previously reported correlation coefficients vary from 0.77 to 0.86. These studies included populations with a wide range of hearing losses, varying from severe to no hearing loss at all.

Based on this relationship, the DIN test could potentially be used as a screening instrument for hearing loss. However, these two studies did not report specifically on a population of elderly subjects, and this is one of the main target groups for hearing screening. It is important to validate the assumed relationship between SRT-in-noise and hearing loss for this particular population with a smartphone, as it may be influenced by general aging, for example, a decline in cognitive skills.

The purpose of this project is to validate a quick, easy-to-use and administer smartphone hearing-in-noise test. The app (called HearMe) can potentially be used to easily and quickly collect hearing-in-noise and speech-in-noise measurements. The smartphone app developed is a hearing-in-noise test that presents the subject with a series of stimuli consisting of a spoken three-digit sequence presented at a varying hearing-to-noise ratio. For each stimulus presentation, the user tap the three-digit sequence. The duration of the app is less than 3 minutes. For this project we will test at least 50 participants with hearing loss and 50 control subjects between the ages of 18-80. The participants will be invited to take the app. The approach for this pilot study is to characterize hearing-in-noise thresholds (also referred to as a speech-reception threshold) as measured by the app in both participant groups, and relate it to the phenotype of each group as a preliminary evaluation of the app as well as a preliminary validation against their routinely collected measurements of hearing function (pure-tone audiometry thresholds).

With this study, the investigators aim to evaluate the developed smartphone HINT/DIN test for its ability to screen the elderly for hearing loss. The investigators hope to examine the relationship between pure-tone thresholds and SRT-in-noise as measured by the HearMe smartphone application.

ELIGIBILITY:
Inclusion Criteria:

* Age-matched (18-100)
* Healthy normal controls with no known hearing loss
* Patients with clinically assessed hearing loss

Exclusion Criteria:

* Complete hearing loss/deafness
* Cognitive decline or dysfunction, dementia

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Standardized Hearing Tests (change in hearing) | Through study completion, an average of 1 year
  Pure-tone audiometry threshold (threshold of hearing relative to frequency)

SECONDARY OUTCOMES:
Quick Hearing Check Questionnaire (change in hearing) | Through study completion, an average of 1 year
  Better Hearing Institute Quick Hearing Check (15 items; score 1-60, higher = better hearing, lower = worse hearing)
Standardized Hearing Loss Questionnaire (change in hearing) | Through study completion, an average of 1 year
  2009 Spatial Hearing Questionnaire (24 items, scored 1-100; higher = better hearing, lower = worse hearing)
Tinnitus Questionnaires (change in hearing) | Through study completion, an average of 1 year
  Tinnitus Activities Questionnaire; Tinnitus Handicap Questionnaire (27 items, scored 1-100%; lower = less effects of tinnitus)

CONTACTS AND LOCATIONS:
Overall Officials: Zarei, Principal Investigator — University of Iowa

IPD SHARING:
Plan to Share IPD: No
There is no intent to make IPD available to other researchers, besides the results published in a peer-reviewed journal publication.

REFERENCES:
- [Background] Ciorba A, Bianchini C, Pelucchi S, Pastore A. The impact of hearing loss on the quality of life of elderly adults. Clin Interv Aging. 2012;7:159-63. doi: 10.2147/CIA.S26059. Epub 2012 Jun 15. PMID 22791988
- [Background] Culling JF, Zhao F, Stephens D. The viability of speech-in-noise audiometric screening using domestic audio equipment. Int J Audiol. 2005 Dec;44(12):691-700. doi: 10.1080/14992020500267017. PMID 16450920
- [Background] Dalton DS, Cruickshanks KJ, Klein BE, Klein R, Wiley TL, Nondahl DM. The impact of hearing loss on quality of life in older adults. Gerontologist. 2003 Oct;43(5):661-8. doi: 10.1093/geront/43.5.661. PMID 14570962
- [Background] Davis A, Smith P, Ferguson M, Stephens D, Gianopoulos I. Acceptability, benefit and costs of early screening for hearing disability: a study of potential screening tests and models. Health Technol Assess. 2007 Oct;11(42):1-294. doi: 10.3310/hta11420. PMID 17927921
- [Background] DePaolis RA, Janota CP, Frank T. Frequency importance functions for words, sentences, and continuous discourse. J Speech Hear Res. 1996 Aug;39(4):714-23. doi: 10.1044/jshr.3904.714. PMID 8844552
- [Background] Grant KW, Walden TC. Understanding excessive SNR loss in hearing-impaired listeners. J Am Acad Audiol. 2013 Apr;24(4):258-73; quiz 337-8. doi: 10.3766/jaaa.24.4.3. PMID 23636208
- [Background] Houtgast T, Festen JM. On the auditory and cognitive functions that may explain an individual's elevation of the speech reception threshold in noise. Int J Audiol. 2008 Jun;47(6):287-95. doi: 10.1080/14992020802127109. PMID 18569101
- [Background] Jansen S, Luts H, Dejonckere P, van Wieringen A, Wouters J. Exploring the sensitivity of speech-in-noise tests for noise-induced hearing loss. Int J Audiol. 2014 Mar;53(3):199-205. doi: 10.3109/14992027.2013.849361. Epub 2013 Nov 18. PMID 24237040
- [Background] Killion MC, Niquette PA, Gudmundsen GI, Revit LJ, Banerjee S. Development of a quick speech-in-noise test for measuring signal-to-noise ratio loss in normal-hearing and hearing-impaired listeners. J Acoust Soc Am. 2004 Oct;116(4 Pt 1):2395-405. doi: 10.1121/1.1784440. PMID 15532670
- [Background] Potgieter JM, Swanepoel de W, Myburgh HC, Hopper TC, Smits C. Development and validation of a smartphone-based digits-in-noise hearing test in South African English. Int J Audiol. 2015 Jul;55(7):405-11. doi: 10.3109/14992027.2016.1172269. Epub 2016 Apr 28. PMID 27121117
- See also: American National Standard, Methods for Calculation of the Speech Intelligibility Index. — http://acousticalsociety.org

DOCUMENTS (1):
  • Study Protocol (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT03429777/Prot_000.pdf